CLINICAL TRIAL: NCT00606424
Title: An Exploratory, Open Label, Single Center Study of [F-18]HX4
Acronym: HX4
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Kathleen Marcozzi Pierce, MA, CNMT, Siemens Molecular Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DHX4000
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 20 mCi dose for a 50 kg individual of [F-18]HX4 — All subjects, normal volunteers and cancer subjects will receive HX4 administered through a previously placed suitably sized angiocatheter or a butterfly needle. Prior to injection, qualified site personnel will assay the dose in the dose calibrator and document the activity of the dose and time of assay. After injection, the line will be flushed with saline (approximately 10 mL).

SUMMARY:
[F-18]HX4 is being developed as a diagnostic radiopharmaceutical for PET imaging. This trial is looking at the safety of [F-18]HX4.

The Sponsor is seeking to determine if [F-18]HX4 may serve as a clinically useful hypoxia marker in diagnostic imaging, allowing the rational application of hypoxia related therapies to those patients most likely to benefit from them.

Tumor hypoxia, a situation where tumor cells have been deprived of oxygen, caused cancer cells to become more resistant to the effects of radiotherapy and chemotherapy.

A non-invasive study characterizing tumor hypoxia would facilitate the development of targeted therapies.

The population to be studied consists of a total of ten (10) adult subjects, including, four normal volunteers and six cancer subjects, the latter with a confirmed diagnosis of head and neck cancer, as defined by the protocol eligibility criteria.

The objectives of this exploratory study are to:

* Gain information on bio-distribution of [F-18]HX4, and to evaluate the PET images of [F-18]HX4 for resolution, signal to background ratio for both intermediate levels of oxygenation, and at extreme levels hypoxia
* Use this eIND in order to obtain the necessary information to file an IND application with the FDA. The information collected under this exploratory study will not be used for diagnostic purposes, to assess the subject's response to therapy, or for clinical management of the subject.
* Begin collection of baseline imaging data
* Collect [F-18]HX4 metabolism data
* Gain information to improve study design and the conduct of future trials

This investigation will be conducted as an exploratory, open-label, non-randomized, uncontrolled, single center, safety study.

The trial is expected to begin subject enrollment in early January 2008 and end subject participation in June 2008.

The duration of an individual subject's participation includes a screening visit, followed by participation in the actual study starting with the day of dosing with imaging sessions lasting several hours, concluding with a next day safety follow-up visit.

Individual doses of [F-18]HX4 shall not exceed 20 mCi. The IP will be administered through a previously placed suitably sized angiocatheter or a butterfly needle. Prior to injection, qualified site personnel will assay the dose. After IP administration several PET imaging series will be acquired. Also, in order to assess major organ function and electrolyte levels, a metabolites analysis will be performed for this study from predose to 90 minutes postdose.

In order to determine the quantity of [F-18]HX4 and labeled metabolites excreted by the kidney,urine will be collected and pooled at the designated intervals after administration of the investigational product. This excretion data will provide supportive information for calculating human dosimetry estimates from PET imaging biodistribution data collected in human subjects.

For cancer subjects, a tissue biopsy will have been taken or be scheduled to be performed. The biopsy sample will be examined for hypoxic biomarker(s) using immunohistochemistry methods.

ELIGIBILITY:
Inclusion Criteria:

Normal Volunteers

* Subject may be male or female and of any race / ethnicity
* Subject is > 18 years old at the time of investigational product administration
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of complying with study procedures
* Subject is capable of communicating with study personnel

Cancer Subjects

* Subject may be male or female and of any race / ethnicity
* Subject is > 18 years old at the time of investigational product administration
* Subject or subject's legally acceptable representative provides written informed consent
* Subject is capable of complying with study procedures
* Subject is capable of communicating with study personnel
* Subject must have histologically confirmed stage III, or IV squamous cell carcinoma of the head and neck whose primary origin was from the oral cavity, oropharynx, hypopharynx, or larynx. Carcinoma must be staged using the American Joint Committee on Cancer (AJCC) staging criteria version 6. Adequate tumor must be amenable to biopsy via outpatient methods
* According to the Karnofsky Performance Status Scale, the subject has a value of ≥ 60% at time of screening
* Subject is scheduled for a clinical FDG PET scan either within 48 hours prior to (with no intervention in between the two scans), or within 48 hours after the investigational [F-18]HX4 PET scan
* Subject must have normal organ and renal function as defined:

  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 x institutional upper limit of normal
  * creatinine within normal institutional limits
  * BUN within normal institutional limits

Exclusion Criteria:

Normal Volunteers

* Subject is younger than 18 years old at the time of investigational product administration
* Female subject is pregnant or nursing--Serum pregnancy test must be negative; test must be completed within 24 hours of dosing or female subject must be either surgically sterilized or post- menopausal, defined as at least one year without menses as reported by the subject
* Subject is unable to remain still for duration of imaging procedure (~40 mins)
* Subject has previously received [F-18]HX4 at any time, or has been involved in an investigative, radioactive research procedure within the past year
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data
* Subject has a history of significant prescription or non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives.

Cancer Subjects

* Subject is younger than 18 years old at the time of investigational product administration
* Female subject is pregnant or has a positive serum pregnancy test
* Subject is unable to remain still for duration of imaging procedure
* Subject has a history of significant renal disease
* Subject has previously received [F-18]HX4 at any time, or any other investigational product in the past thirty days.
* Subject has been involved in an investigative, radioactive research procedure within the past year
* Inadequate tumor sites or volume to allow for biopsy
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete and good quality data
* Subject has a history of significant prescription or non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety will be the outcome demonstrated in this clinical trial through analyses of adverse events in subjects who receive study drug. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yu, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Michael Yu, MD, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Doss M, Zhang JJ, Belanger MJ, Stubbs JB, Hostetler ED, Alpaugh K, Kolb HC, Yu JQ. Biodistribution and radiation dosimetry of the hypoxia marker 18F-HX4 in monkeys and humans determined by using whole-body PET/CT. Nucl Med Commun. 2010 Dec;31(12):1016-24. doi: 10.1097/MNM.0b013e3283407950. PMID 20948452